CLINICAL TRIAL: NCT07083375
Title: A Phase II Clinical Trial of Iparomlimab and Tuvonralimab in Combination With Bevacizumab and Platinum-based Chemotherapy in Previously Untreated Patients With Extensive-stage Small Cell Lung Cancer.
Brief Title: A Phase II Study of QL1706 With Anti-angiogenesis Therapy and Chemotherapy in Extensive-stage Small Cell Lung Cancer.
Acronym: QL1706
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhijie Wang (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Hebei Medical University Fourth Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Renmin Hospital of Wuhan University (Other); Wuhan TongJi Hospital (Other); Peking University People's Hospital (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhijie Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5301
Record Dates: First submitted 2025-07-07; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Extensive Small Cell Lung Cancer
Keywords: QL1706; Extensive Small Cell Lung Cancer; combination therapy; first line therapy
MeSH Terms: interventions — Bevacizumab; Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined treatment group (Experimental): This study investigates a novel four-drug first-line treatment for extensive-stage small cell lung cancer (ES-SCLC), combining QL1706-a bifunctional antibody targeting both PD-1 and CTLA-4-with bevacizumab (anti-VEGF) and platinum-based chemotherapy (etoposide + cisplatin or carboplatin). QL1706 is uniquely engineered to provide dual checkpoint inhibition with reduced CTLA-4 exposure, potentially enhancing efficacy while limiting immune-related toxicity. Bevacizumab adds antiangiogenic activity, aiming to improve immune infiltration and drug delivery. This synergistic approach integrates immunotherapy, antiangiogenesis, and cytotoxic agents to overcome resistance and extend survival. All patients receive dual-agent maintenance (QL1706 + bevacizumab) post-induction. No prior studies have evaluated this specific combination in ES-SCLC.
  Interventions: Drug: QL1706 , bevacizumab, etoposide , cisplatin or carboplatin

INTERVENTIONS:
Drug: QL1706 , bevacizumab, etoposide , cisplatin or carboplatin — Participants will receive QL1706 (5 mg/kg, IV, day 1), bevacizumab (7.5 mg/kg, IV, day 1), etoposide (100 mg/m², IV, days 1-3), plus either cisplatin (75 mg/m² split over days 1-2, IV) or carboplatin (AUC=5, IV, day 1) every 21 days for 4-6 cycles. Dose adjustments may be made based on clinical judgment. Patients who do not experience disease progression or intolerable toxicity will proceed to maintenance therapy with QL1706 (5 mg/kg, IV, day 1) and bevacizumab (7.5 mg/kg, IV, day 1) every 21 days, continued until disease progression, unacceptable toxicity, consent withdrawal, investigator decision, loss to follow-up, death, or other protocol-defined criteria. All participants will receive dual-agent maintenance therapy.

SUMMARY:
This single-arm, open-label, Phase II study assesses first-line QL1706 + bevacizumab (anti-VEGF) + platinum/etoposide chemotherapy to treat naïve ES-SCLC patients.The main questions it aims to answer are:

Evaluate efficacy and safety of this quadruplet regimen in ES-SCLC Explore correlations between tumor biomarkers and treatment efficacy

Participants will:

Histologically or cytologically confirmed, treatment-naïve extensive-stage small cell lung cancer (ES-SCLC).

Willing to provide archived or fresh tumor tissue samples. If unavailable, enrollment may proceed per investigator assessment.

At least one measurable lesion per RECIST v1.1

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is a highly aggressive malignancy, accounting for 13-15% of all lung cancers. Approximately two-thirds of patients present with distant metastases at diagnosis, defined as extensive-stage SCLC (ES-SCLC). Prognosis remains poor, with median overall survival (mOS) of 12-15 months despite standard first-line chemotherapy using etoposide plus cisplatin/carboplatin (EP/EC), which offers limited benefit (mOS ~10 months; median progression-free survival [mPFS] ~5 months).

Immune checkpoint inhibitors (ICIs) have improved outcomes modestly. IMpower133, KEYNOTE-604, RATIONALE-312, and EXTENTORCH trials confirmed the benefit of adding PD-1/PD-L1 inhibitors to chemotherapy, but the survival plateau remains. Dual immune checkpoint blockade strategies, including PD-1/PD-L1 with CTLA-4 inhibitors, have not significantly improved outcomes and pose higher toxicity, as seen in CASPIAN and CheckMate451 studies.

Antiangiogenic therapy offers another promising direction. Studies such as SALUTE, ACTION-2, and BEAT-SC have explored bevacizumab or anlotinib combined with chemo-immunotherapy, showing potential survival gains. Notably, the ETER701 study using a four-drug combination achieved mOS of 19.3 months, although with increased adverse events.

QL1706 (Aito combination antibody) is a novel bifunctional antibody targeting PD-1 and CTLA-4 in a 2:1 fixed ratio, designed to optimize synergy while reducing CTLA-4 toxicity. Approved in 2024, it has demonstrated efficacy and tolerability in multiple solid tumors. In NSCLC, QL1706 combined with chemotherapy and antiangiogenic therapy showed mPFS up to 8.5 months and mOS of 26.5 months.

To date, no clinical data exist for QL1706 combined with antiangiogenic therapy and chemotherapy in ES-SCLC. A phase II, open-label, single-arm clinical trial is proposed to evaluate its efficacy and safety as first-line treatment. This study aims to explore a new therapeutic strategy to overcome the current survival limitations in ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the study:

1. Signed written informed consent and willingness to comply with study procedures.
2. Age ≥18 years.
3. Estimated life expectancy ≥3 months.
4. ECOG performance status of 0 or 1.
5. Histologically or cytologically confirmed, treatment-naïve extensive-stage small cell lung cancer (ES-SCLC).
6. Willing to provide archived or fresh tumor tissue samples. If unavailable, enrollment may proceed per investigator assessment.
7. At least one measurable lesion per RECIST v1.1.
8. Fully understands and voluntarily participates in the study.
9. Adequate organ function as defined below:

   * Absolute neutrophil count ≥1.5 × 10⁹/L
   * Platelets ≥100 × 10⁹/L
   * Hemoglobin ≥90 g/L (without transfusion in prior 14 days)
   * Serum creatinine ≤1× ULN or creatinine clearance >50 mL/min (Cockcroft-Gault)
   * AST and ALT ≤2.5× ULN (≤5× ULN with liver metastases)
   * Total bilirubin ≤1.5× ULN (except Gilbert's syndrome <51.3 µmol/L)
   * TSH, FT3, FT4 within ±10% of normal limits

Exclusion Criteria:

1. Prior chemotherapy, immunotherapy, targeted therapy, or radiotherapy.
2. Histologic or cytologic evidence of non-small cell or mixed small cell/non-small cell carcinoma.
3. Symptomatic brain metastases or leptomeningeal disease.
4. Active or suspected autoimmune disease, except for stable vitiligo, type 1 diabetes, hypothyroidism requiring only hormone replacement, or conditions not expected to recur.
5. Evidence or history of active pulmonary tuberculosis (TB), including treated TB within the past year.
6. Concomitant condition requiring systemic corticosteroids or other immunosuppressive therapy.
7. Pregnant or breastfeeding females.
8. Symptomatic interstitial lung disease or suspected drug-related pneumonitis.
9. Positive for HIV antibodies, active HBV (HBsAg+ with HBV DNA >10³ copies/mL), or active HCV infection (HCV-Ab+ with detectable RNA).
10. History of significant neurological or psychiatric disorders (e.g., dementia, depression, epilepsy, bipolar disorder).
11. Participation in another investigational drug study within 4 weeks prior to randomization.
12. Use of anti-tumor traditional Chinese medicine within 2 weeks prior to first study dose.
13. History of other malignancies within 2 years, except for cured non-melanoma skin cancers or certain in situ carcinomas.
14. Clinically significant cardiovascular or cerebrovascular disease (e.g., NYHA class ≥2 heart failure, recent myocardial infarction or stroke within 6 months).
15. History of thromboembolic events (e.g., DVT, PE, arterial thrombosis) within 6 months, except catheter-related thrombosis.
16. Live vaccination within 28 days before randomization or planned during the study.
17. Major surgery or significant trauma within 4 weeks prior to treatment initiation.
18. Conditions affecting drug absorption (e.g., severe vomiting, GI obstruction, active GI bleeding or perforation).
19. Active, uncontrolled bacterial, viral, or fungal infections despite appropriate treatment.
20. Known hypersensitivity to any study drug or excipients.
21. Any other condition deemed unsuitable by the investigator due to safety or compliance concerns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to the end of monitoring at 2 years.
  PFS is defined as the time from the first dose of study treatment to the first documentation of disease progression according to RECIST v1.1 (as assessed by investigators) or death from any cause, whichever occurs first. Subjects who are alive without progression at the time of analysis will be censored at the date of the last tumor assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to the end of monitoring at 2 years.
  OS is defined as the time from the first dose of study treatment to death from any cause. Subjects who are alive at the time of analysis will be censored at the date of last follow-up.
Objective Response Rate (ORR) | From enrollment to the end of monitoring at 2 years.
  ORR is defined as the proportion of subjects who achieve a complete response (CR) or partial response (PR) as per RECIST v1.1.
Duration of Response (DoR) | From enrollment to the end of monitoring at 2 years.
  DoR is defined as the time from the first documentation of CR or PR to the first documentation of disease progression or death.
Disease Control Rate (DCR) | From enrollment to the end of monitoring at 2 years.
  DCR is defined as the proportion of subjects who achieve CR, PR, or stable disease (SD) as their best overall response.
The incidence of adverse events | From enrollment to the end of monitoring at 2 years
  Incidence, nature, and severity of adverse events (AEs), graded according to NCI-CTCAE v5.0, including immune-related AEs and serious AEs.

OTHER OUTCOMES:
Immune-Related Adverse Events (irAEs) | From enrollment to the end of monitoring at 2 years
  Occurrence and grade of immune-related adverse events as defined by pre-specified criteria, including rash, colitis, hepatitis, endocrinopathies, and pneumonitis.
Biomarker Analysis | From enrollment to the end of monitoring at 2 years
  Tumor tissues were detected for PD-L1 using IHC. Potential biomarkers such as CD3+ and CD8+ were detected in peripheral blood.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing 100021, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Deng P, Kong T, Zhang B, Qian F, Dong Y, Chen Y, Chen L, Liu D, Zhang Y, Yang H, Han B. Safety and efficacy of anlotinib in combination with standard chemotherapy as first-line treatment for extensive-stage small cell lung cancer: A multi-center, prospective study (ACTION-2). Lung Cancer. 2022 Nov;173:43-48. doi: 10.1016/j.lungcan.2022.09.003. Epub 2022 Sep 8. PMID 36116169
- [Background] Reck M, Luft A, Szczesna A, Havel L, Kim SW, Akerley W, Pietanza MC, Wu YL, Zielinski C, Thomas M, Felip E, Gold K, Horn L, Aerts J, Nakagawa K, Lorigan P, Pieters A, Kong Sanchez T, Fairchild J, Spigel D. Phase III Randomized Trial of Ipilimumab Plus Etoposide and Platinum Versus Placebo Plus Etoposide and Platinum in Extensive-Stage Small-Cell Lung Cancer. J Clin Oncol. 2016 Nov 1;34(31):3740-3748. doi: 10.1200/JCO.2016.67.6601. PMID 27458307
- [Background] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938
- [Background] Hong MMY, Maleki Vareki S. Addressing the Elephant in the Immunotherapy Room: Effector T-Cell Priming versus Depletion of Regulatory T-Cells by Anti-CTLA-4 Therapy. Cancers (Basel). 2022 Mar 20;14(6):1580. doi: 10.3390/cancers14061580. PMID 35326731
- [Background] Cheng Y, Chen J, Zhang W, Xie C, Hu Q, Zhou N, Huang C, Wei S, Sun H, Li X, Yu Y, Lai J, Yang H, Fang H, Chen H, Zhang P, Gu K, Wang Q, Shi J, Yi T, Xu X, Ye X, Wang D, Xie C, Liu C, Zheng Y, Lin D, Zhuang W, Lu P, Yu G, Li J, Gu Y, Li B, Wu R, Jiang O, Wang Z, Wu G, Lin H, Zhong D, Xu Y, Shu Y, Wu D, Chen X, Wang J, Wang M, Yang R. Benmelstobart, anlotinib and chemotherapy in extensive-stage small-cell lung cancer: a randomized phase 3 trial. Nat Med. 2024 Oct;30(10):2967-2976. doi: 10.1038/s41591-024-03132-1. Epub 2024 Jul 11. PMID 38992123
- [Background] Lamberti G, Rihawi K, Mazzoni F, Riccardi F, Follador A, Tiseo M, Frassoldati A, Colantonio I, Bonetti A, Genova C, Giardina D, Bertolini F, Cinieri S, Pasello G, Brighenti M, Andrini E, Tognetto M, Boni L, Ardizzoni A; GOIRC group. Carboplatin, etoposide, atezolizumab, and bevacizumab in the first-line treatment of patients with extensive stage small-cell lung cancer: the GOIRC-01-2019 CeLEBrATE study. J Immunother Cancer. 2025 May 7;13(5):e010694. doi: 10.1136/jitc-2024-010694. PMID 40341031
- [Background] Spigel DR, Townley PM, Waterhouse DM, Fang L, Adiguzel I, Huang JE, Karlin DA, Faoro L, Scappaticci FA, Socinski MA. Randomized phase II study of bevacizumab in combination with chemotherapy in previously untreated extensive-stage small-cell lung cancer: results from the SALUTE trial. J Clin Oncol. 2011 Jun 1;29(16):2215-22. doi: 10.1200/JCO.2010.29.3423. Epub 2011 Apr 18. PMID 21502556
- [Background] Xie M, Vuko M, Rodriguez-Canales J, Zimmermann J, Schick M, O'Brien C, Paz-Ares L, Goldman JW, Garassino MC, Gay CM, Heymach JV, Jiang H, Barrett JC, Stewart RA, Lai Z, Byers LA, Rudin CM, Shrestha Y. Molecular classification and biomarkers of outcome with immunotherapy in extensive-stage small-cell lung cancer: analyses of the CASPIAN phase 3 study. Mol Cancer. 2024 May 30;23(1):115. doi: 10.1186/s12943-024-02014-x. PMID 38811992
- [Background] Thomas BL, Tucker AS, Ferguson C, Qiu M, Rubenstein JL, Sharpe PT. Molecular control of odontogenic patterning: positional dependent initiation and morphogenesis. Eur J Oral Sci. 1998 Jan;106 Suppl 1:44-7. doi: 10.1111/j.1600-0722.1998.tb02152.x. PMID 9541202
- [Background] Cheng Y, Fan Y, Zhao Y, Huang D, Li X, Zhang P, Kang M, Yang N, Zhong D, Wang Z, Yu Y, Zhang Y, Zhao J, Qin T, Chen C, Leaw S, Zheng W, Song Y; RATIONALE-312 Study Group. Tislelizumab Plus Platinum and Etoposide Versus Placebo Plus Platinum and Etoposide as First-Line Treatment for Extensive-Stage SCLC (RATIONALE-312): A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Phase 3 Clinical Trial. J Thorac Oncol. 2024 Jul;19(7):1073-1085. doi: 10.1016/j.jtho.2024.03.008. Epub 2024 Mar 7. PMID 38460751
- [Background] Rudin CM, Awad MM, Navarro A, Gottfried M, Peters S, Csoszi T, Cheema PK, Rodriguez-Abreu D, Wollner M, Yang JC, Mazieres J, Orlandi FJ, Luft A, Gumus M, Kato T, Kalemkerian GP, Luo Y, Ebiana V, Pietanza MC, Kim HR; KEYNOTE-604 Investigators. Pembrolizumab or Placebo Plus Etoposide and Platinum as First-Line Therapy for Extensive-Stage Small-Cell Lung Cancer: Randomized, Double-Blind, Phase III KEYNOTE-604 Study. J Clin Oncol. 2020 Jul 20;38(21):2369-2379. doi: 10.1200/JCO.20.00793. Epub 2020 May 29. PMID 32468956
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Sokol R, Pluta P. ENDOPARASITES IN WESTERN CAPERCAILLIES (TETRAO UROGALLUS) AND BLACK GROUSE (TETRAO TETRIX) KEPT IN VARIOUS TYPES OF AVIARIES. J Wildl Dis. 2022 Jan 1;58(1):114-121. doi: 10.7589/JWD-D-21-00017. PMID 34714912
- [Background] Han S, Gelernter J, Kranzler HR, Yang BZ. Ordered subset linkage analysis based on admixture proportion identifies new linkage evidence for alcohol dependence in African-Americans. Hum Genet. 2013 Apr;132(4):397-403. doi: 10.1007/s00439-012-1255-2. Epub 2012 Dec 13. PMID 23239122
- [Background] Gazdar AF, Bunn PA, Minna JD. Small-cell lung cancer: what we know, what we need to know and the path forward. Nat Rev Cancer. 2017 Nov 10;17(12):765. doi: 10.1038/nrc.2017.106. Online ahead of print. PMID 29123245
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204